CLINICAL TRIAL: NCT03048357
Title: Effectiveness of the Freedom Bed, Automatic Continuous Lateral Rotation Therapy System as Compared to a Standard Hospital Mattress With Manual Caregiver Turning Every 2 Hours for Prevention of Pressure Injuries in Persons With Limited Mobility Due to Traumatic Brain Injury and/or Spinal Cord Injury.
Brief Title: Effectiveness of Freedom Bed Compared to Manual Turning in Prevention of Pressure Injuries in Persons With Limited Mobility Due to Traumatic Brain Injury and/or Spinal Cord Injury.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northeast Center for Rehabilitation and Brain Injury (Other)
Collaborators: Probed Medical USA (Unknown)
Responsible Party: Principal Investigator, Annmarie Belfiglio, Occupational Therapy Coordinator, Northeast Center for Rehabilitation and Brain Injury
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 2
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Freedom Bed (Active Comparator): Freedom Bed Continuous Lateral Rotation Therapy System
  Interventions: Device: Freedom Bed
- Standard Hospital Bed & Protocol (Other): Standard Hospital Bed with manual caregiver re-positioning every 2 hours
  Interventions: Other: Standard hospital bed

INTERVENTIONS:
Device: Freedom Bed — Fully Integrated Lateral Rotation Bed System that automatically turns the patient to a specific angle in degrees between from 15-25 with dwell times between 1-120 minutes.
  Arms: Freedom Bed
Other: Standard hospital bed — Caregiver turning patients to one side then the other every 2 hours for pressure relief over bony prominence's.
  Arms: Standard Hospital Bed & Protocol

SUMMARY:
Observational comparison on Incidence of Pressure Injury between the Freedom Bed Automated Continuous lateral Rotation Therapy System and Manual Caregiver Re-positioning every 2 hours on a standard Hospital Bed.

DETAILED DESCRIPTION:
This study will include 8 vent dependent subjects with comparable diagnoses and nutritional levels. Of the subjects selected, 4 subjects will be placed on Freedom Beds and 4 will be placed on standard hospital beds for a period not less than 6 months. A waiver of informed consent is required prior to bed placement and data collection. Consented subjects will have primary and secondary diagnosis recorded, pressure mapping in supine 30-degree elevation, assessment of ventilator / oxygen support measured, oxygenation levels, nutrition levels, and estimated cardiac condition. Subjects will receive daily skin assessments and treatment as prescribed by the attending physician with weekly measurements and reporting of values. Subjects will continue until they reach one of the study endpoints: 1) discharge from the vent unit, or 2) withdrawal of informed consent, or 3) completion of the 6-month study.

Subjects placed on the Freedom Bed will be automatically turned in accordance with positions determined as optimal by initial pressure mapping and approved by the attending physician. All programmable turning angles, dwell times, head and leg elevations must be "dialed in" within a week of the study beginning. Any modification to the program during the study must be approved by the care team and documented accordingly.

Subjects placed on standard hospital bed will require manual re-positioning every 2 hours. All turning and/or re-positioning must be timed and documented.

Subjects who experience either development of pressure injuries, or worsening of their skin condition to the point a specialty bed is required will be deemed a test failure.

The primary and secondary outcome measures documented on each subject throughout the week will be collected by the Clinical Research Coordinator (CRC) on a weekly basis and submitted to the Principal Investigator. The weekly reports will then be consolidated by the CRC into a monthly report and submitted to the Institutional Review Board (IRB), Principal Investigators (PI) and Supervising Authorities (SA) for review.

ELIGIBILITY:
Inclusion Criteria:

Subjects or their legal representative able to provide written consent for study Must be rated between 6-12 on the Baden Scale Must be immobile and unable to preposition themselves. Must be within weight range of designated support surface.

Exclusion Criteria:

Subjects with unstable spinal fractures. Subjects with significant involuntary spasms. Subjects with severe scoliosis. A user must be able to lie in a partial back lying position.

Subjects considered morbidly obese.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Pressure Injury | 12 months

SECONDARY OUTCOMES:
Incidence of Pneumonia | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine McCalister, M.S., Study Director — Director Of Therapy, Northeast Center

IPD SHARING:
Plan to Share IPD: No